CLINICAL TRIAL: NCT00687193
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Confirm Dose Responsiveness Following 12 Weeks Of The Administration Of CP-690,550 (5 Doses) Or Placebo In Subjects With Active Rheumatoid Arthritis Inadequately Responding To At Least 1 DMARD
Brief Title: Comparison Of 5 CP-690,550 Doses Vs. Placebo, For The Treatment Of Rheumatoid Arthritis In Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921040
Record Dates: First submitted 2008-05-22; First posted 2008-05-30 (Estimated); Results first posted 2012-12-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Phase 2 monotherapy in Japan
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CP-690,550, 10mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 15mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 1mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 3mg (Experimental)
  Interventions: Drug: CP-690,550
- CP-690,550, 5mg (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Placebo — Placebo BID, 3 blinded tablets administered BID for 12 weeks
  Arms: Placebo
Drug: CP-690,550 — 10mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 10mg
Drug: CP-690,550 — 15mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 15mg
Drug: CP-690,550 — 1mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 1mg
Drug: CP-690,550 — 3mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 3mg
Drug: CP-690,550 — 5mg BID, 3 blinded tablets administered BID for 12 weeks
  Arms: CP-690,550, 5mg

SUMMARY:
To evaluate the dose-response relationship of 5 dose of CP-690,550, compared to placebo for the treatment of signs and symptoms in patients with active RA who failed an adequate trial of therapy with at least 1 DMARD in a 12-week therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have failed an adequate trial of therapy with at least 1 DMARD due to lack of efficacy or toxicity.

Exclusion Criteria:

* Current therapy with any DMARD

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- Japan (40):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Narashino, Chiba
  - Pfizer Investigational Site, Yotukaidou, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Iiduka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Kurume, Fukuoka
  - Pfizer Investigational Site, Sawara-ku, Fukuoka
  - Pfizer Investigational Site, Fukushima, Fukushima
  - Pfizer Investigational Site, Takasaki, Gunma
  - Pfizer Investigational Site, Higashihiroshima, Hiroshima
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Asahikawa, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Nishinomiya, Hyōgo
  - Pfizer Investigational Site, Tsukuba, Ibaraki
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Koushi, Kumamoto
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Nagasaki, Nagasaki
  - Pfizer Investigational Site, Ohmura, Nagasaki
  - Pfizer Investigational Site, Sasebo, Nagasaki
  - Pfizer Investigational Site, Kashihara, Nara
  - Pfizer Investigational Site, Ōita, Oita Prefecture
  - Pfizer Investigational Site, Kawachi-Nagano, Osaka
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Ureshino-shi, Saga-ken
  - Pfizer Investigational Site, Kawagoe-shi, Saitama
  - Pfizer Investigational Site, Kitamoto, Saitama
  - Pfizer Investigational Site, Saitama, Saitama
  - Pfizer Investigational Site, Arakawa-ku, Tokyo
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Musashimurayama-shi, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinjyuku-ku, Tokyo
  - Pfizer Investigational Site, Takaoka, Toyama

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Charles-Schoeman C, Hyde C, Guan S, Parikh N, Wang J, Shahbazian A, Stockert L, Andrews J. Relationship Between Paraoxonase-1 Genotype and Activity, and Major Adverse Cardiovascular Events and Malignancies in Patients With Rheumatoid Arthritis Receiving Tofacitinib. J Rheumatol. 2023 Jul 15:jrheum.2023-0112. doi: 10.3899/jrheum.2023-0112. Online ahead of print. PMID 37453736
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Suzuki M, Shoji S, Miyoshi S, Krishnaswami S. Model-Based Comparison of Dose-Response Profiles of Tofacitinib in Japanese Versus Western Rheumatoid Arthritis Patients. J Clin Pharmacol. 2020 Feb;60(2):198-208. doi: 10.1002/jcph.1514. Epub 2019 Sep 12. PMID 31512746
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Charles-Schoeman C, Burmester G, Nash P, Zerbini CA, Soma K, Kwok K, Hendrikx T, Bananis E, Fleischmann R. Efficacy and safety of tofacitinib following inadequate response to conventional synthetic or biological disease-modifying antirheumatic drugs. Ann Rheum Dis. 2016 Jul;75(7):1293-301. doi: 10.1136/annrheumdis-2014-207178. Epub 2015 Aug 14. PMID 26275429
- [Derived] Tanaka Y, Takeuchi T, Yamanaka H, Nakamura H, Toyoizumi S, Zwillich S. Efficacy and safety of tofacitinib as monotherapy in Japanese patients with active rheumatoid arthritis: a 12-week, randomized, phase 2 study. Mod Rheumatol. 2015 Jul;25(4):514-21. doi: 10.3109/14397595.2014.995875. PMID 25496464
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921040&StudyName=Comparison%20Of%205%20CP-690%2C550%20Doses%20Vs.%20Placebo%2C%20For%20The%20Treatment%20Of%20Rheumatoid%20Arthritis%20In%20Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 1 mg: Participants were administered 1 milligram (mg) of CP-690,550 orally twice daily for 12 weeks.
- CP-690,550 3 mg: Participants were administered 3 mg of CP-690,550 orally twice daily for 12 weeks.
- CP-690,550 5 mg: Participants were administered 5 mg of CP-690,550 orally twice daily for 12 weeks.
- CP-690,550 10 mg: Participants were administered 10 mg of CP-690,550 orally twice daily for 12 weeks.
- CP-690,550 15 mg: Participants were administered 15 mg of CP-690,550 orally twice daily for 12 weeks.
- Placebo: Participants were administered placebo tablet matched to CP-690,550 orally twice daily for 12 weeks.
Period: Overall Study
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Started | 53 | 53 | 52 | 53 | 54 | 52 (One participant withdrew after randomization but prior to treatment.)
Completed | 51 | 49 | 50 | 49 | 52 | 48
Not Completed | 2 | 4 | 2 | 4 | 2 | 4
Not completed — Adverse Event | 0 | 1 | 2 | 3 | 0 | 2
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 2 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52 | 317
Age, Customized [Number; unit: Participants]
  < 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 8 | 11 | 13 | 9 | 12 | 14 | 67
  Between 45 and 64 years | 39 | 33 | 31 | 32 | 30 | 29 | 194
  >= 65 years | 6 | 9 | 8 | 12 | 12 | 9 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 47 | 44 | 44 | 44 | 43 | 264
  Male | 11 | 6 | 8 | 9 | 10 | 9 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in painful and tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 12
Population: The full analysis set included all participants who were randomized to the study and received at least 1 dose of study medication. Missing values were handled using the Last Observation Carried Forward (LOCF) method.
Measure: Number; unit: participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
participants | 20 | 36 | 38 | 45 | 49 | 8

2. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Weeks 2, 4 and 8
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in painful and tender joint count; >= 20% improvement in swollen joint count; and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP)at each visit.
Time Frame: Week 2, 4, and 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
participants
  Week 2 (LOCF) | 10 | 18 | 18 | 35 | 29 | 3
  Week 4 (LOCF) | 19 | 25 | 32 | 43 | 42 | 5
  Week 8 (LOCF) | 20 | 33 | 35 | 46 | 47 | 6

3. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: greater than or equal to (>=) 50 percent (%) improvement in painful and tender joint count; >= 50% improvement in swollen joint count; and >= 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Time Frame: Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 54 | 52
participants
  Week 2 (LOCF) | 1 | 5 | 6 | 17 | 12 | 0
  Week 4 (LOCF) | 5 | 12 | 15 | 29 | 25 | 1
  Week 8 (LOCF) | 6 | 20 | 23 | 33 | 36 | 1
  Week 12 (LOCF) | 7 | 14 | 24 | 37 | 39 | 4

4. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: greater than or equal to (>=) 70 percent (%) improvement in painful and tender joint count; >= 70% improvement in swollen joint count; and >= 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Time Frame: Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
participants
  Week 2 (LOCF) | 0 | 0 | 1 | 5 | 4 | 0
  Week 4 (LOCF) | 1 | 2 | 9 | 14 | 9 | 0
  Week 8 (LOCF) | 3 | 7 | 13 | 20 | 22 | 1
  Week 12 (LOCF) | 4 | 7 | 14 | 26 | 28 | 1

5. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 90% (ACR90) Response
Description: ACR90 response: greater than or equal to (>=) 90 percent (%) improvement in painful and tender joint count; >= 90% improvement in swollen joint count; and >= 90% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP) at each visit.
Time Frame: Week 2, 4, 8 and 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
participants
  Week 2 (LOCF) | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 (LOCF) | 0 | 0 | 0 | 2 | 3 | 0
  Week 8 (LOCF) | 0 | 0 | 3 | 7 | 5 | 0
  Week 12 (LOCF) | 0 | 0 | 2 | 8 | 6 | 0

6. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count Using C-reactive Protein [DAS28-3(CRP)]
Description: The DAS28-3 (CRP) score is a measure of the perticipant's disease activity. It is based on the painful and tender joint count (28 joints), swollen joint count (28 joints) and CRP. DAS28-3 (CRP) scores range from 0 - 10; higher scores indicated greater affectation due to disease activity.
  Change = value at observation minus value at baseline
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: The full analysis set included all participants who were randomized to the study and received at least 1 dose of study medication. Missing values were not imputed.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- CP-690,550 1 mg: Participants were administered 1 milligram (mg) of CP-690,550 orally twice daily for 12 weeks. Missing values were not imputed.
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -0.56 (0.13) | -1.03 (0.13) | -1.01 (0.13) | -1.65 (0.13) | -1.63 (0.13) | -0.20 (0.13)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -0.82 (0.13) | -1.29 (0.13) | -1.65 (0.13) | -2.33 (0.13) | -2.14 (0.13) | -0.23 (0.13)
  Week 8 (n=51, 51, 51, 52, 52, 50) | -0.98 (0.13) | -1.63 (0.13) | -1.95 (0.13) | -2.62 (0.13) | -2.55 (0.13) | -0.15 (0.13)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -1.09 (0.13) | -1.71 (0.13) | -2.02 (0.13) | -2.81 (0.13) | -2.70 (0.13) | -0.12 (0.13)

7. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count Using Erythrocyte Sedimentation Rate [DAS28-4(ESR)]
Description: The DAS28-4 (ESR) score is a measure of the participant's disease activity. It is based on the painful and tender joint count (28 joints), swollen joint count (28 joints), participant's global assessment of disease activity (mm), and ESR. DAS28-4(ESR) scores range from 0 - 10; higher scores indicated greater affectation due to disease activity.
  Change = score at observation minus score at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=52, 53, 50, 52, 54, 52) | -0.52 (0.15) | -0.93 (0.14) | -1.00 (0.15) | -1.66 (0.15) | -1.58 (0.14) | -0.25 (0.15)
  Week 4 (n=52, 51, 51, 52, 52, 51) | -0.79 (0.15) | -1.32 (0.15) | -1.69 (0.15) | -2.42 (0.15) | -2.31 (0.14) | -0.23 (0.15)
  Week 8 (n=51, 50, 51, 52, 52, 50) | -1.03 (0.15) | -1.68 (0.15) | -2.05 (0.15) | -2.92 (0.15) | -2.87 (0.14) | -0.12 (0.15)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -1.10 (0.15) | -1.74 (0.15) | -2.20 (0.15) | -3.05 (0.15) | -2.98 (0.14) | -0.10 (0.15)

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
  Change = score at observation minus score at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -0.10 (0.06) | -0.15 (0.06) | -0.28 (0.06) | -0.39 (0.06) | -0.40 (0.06) | 0.06 (0.06)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -0.07 (0.06) | -0.25 (0.06) | -0.38 (0.06) | -0.54 (0.06) | -0.51 (0.06) | 0.03 (0.06)
  Week 8 (n=51, 50, 51, 52, 52, 50) | -0.17 (0.06) | -0.36 (0.06) | -0.49 (0.06) | -0.59 (0.06) | -0.63 (0.06) | 0.18 (0.06)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -0.19 (0.06) | -0.38 (0.06) | -0.55 (0.06) | -0.67 (0.06) | -0.68 (0.06) | 0.18 (0.06)

9. Secondary Outcome: Change From Baseline in Painful and Tender Joint Counts
Description: Number of tender joints was determined by examining 68 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1. A negative value in change from baseline indicates an improvement. Change = value at observation minus value at baseline.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -4.14 (0.98) | -5.13 (0.97) | -5.29 (0.99) | -8.48 (0.98) | -7.73 (0.96) | -2.03 (0.98)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -5.92 (0.98) | -6.95 (0.98) | -8.41 (0.99) | -11.35 (0.98) | -10.41 (0.97) | -1.12 (0.98)
  Week 8 (n=51, 51, 51, 52, 52, 50) | -6.27 (0.98) | -8.80 (0.98) | -9.65 (0.99) | -12.89 (0.98) | -12.16 (0.97) | -0.49 (0.99)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -7.05 (0.98) | -10.01 (0.99) | -10.08 (1.00) | -13.67 (0.99) | -12.81 (0.97) | -0.67 (1.00)

10. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC)
Description: Number of swollen joints was determined by examination of 66 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1. A negative value in change from baseline indicates an improvement. Change = value at observation minus value at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -3.19 (0.69) | -3.85 (0.68) | -2.58 (0.70) | -6.93 (0.69) | -5.95 (0.68) | -1.58 (0.69)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -4.57 (0.69) | -6.10 (0.69) | -6.15 (0.70) | -8.85 (0.69) | -8.15 (0.68) | -1.87 (0.69)
  Week 8 (n=51, 51, 51, 52, 52, 50) | -5.25 (0.69) | -7.08 (0.69) | -7.15 (0.70) | -10.04 (0.69) | -10.52 (0.68) | -1.70 (0.70)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -5.76 (0.69) | -7.94 (0.70) | -7.75 (0.70) | -10.44 (0.70) | -10.73 (0.68) | -1.29 (0.70)

11. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain
Description: Change from Baseline in Patient's Assessment of Arthritis Pain -VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) was computed as Week 2, 4, 8 or 12 values minus baseline value. A negative value in change from baseline indicates an improvement.
  Change = value at observation minus value at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -8.63 (2.94) | -16.70 (2.94) | -19.13 (3.01) | -29.03 (2.97) | -26.45 (2.92) | -1.46 (2.98)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -12.97 (2.96) | -21.19 (2.98) | -26.06 (3.01) | -36.65 (2.97) | -35.16 (2.95) | -2.73 (2.98)
  Week 8 (n=51, 50, 51, 52, 52, 50) | -17.57 (2.97) | -26.15 (2.99) | -30.37 (3.01) | -41.84 (2.97) | -43.08 (2.95) | 1.65 (3.01)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -18.38 (2.97) | -22.33 (3.00) | -34.37 (3.02) | -42.91 (3.01) | -43.79 (2.95) | -1.06 (3.03)

12. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using a 0 - 100 mm Visual Analog Scale where 0 = very well and 100 = very poorly. Change = score at observation minus score at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -7.66 (2.96) | -15.25 (2.97) | -20.32 (3.04) | -27.06 (2.99) | -26.80 (2.94) | -1.73 (3.00)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -11.22 (2.98) | -23.17 (3.00) | -27.03 (3.04) | -36.64 (2.99) | -35.96 (2.97) | -3.31 (3.00)
  Week 8 (n=51, 50, 51, 52, 52, 50) | -16.66 (2.99) | -24.60 (3.01) | -28.78 (3.04) | -41.97 (2.99) | -41.13 (2.97) | 0.79 (3.03)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -16.29 (2.99) | -20.91 (3.03) | -34.59 (3.05) | -43.55 (3.03) | -41.86 (2.97) | -1.02 (3.05)

13. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity; very good and 100 mm = worst disease activity; very poor. Change = score at observation minus score at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
Units on a scale
  Week 2 (n=53, 53, 51, 52, 54, 52) | -13.97 (2.64) | -15.86 (2.63) | -18.10 (2.70) | -31.59 (2.66) | -25.93 (2.61) | -6.09 (2.66)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -23.31 (2.65) | -26.22 (2.67) | -30.45 (2.70) | -41.21 (2.66) | -37.07 (2.64) | -9.70 (2.66)
  Week 8 (n=51, 51, 51, 52, 52, 50) | -21.99 (2.66) | -32.04 (2.67) | -36.92 (2.70) | -45.98 (2.66) | -44.66 (2.64) | -6.84 (2.69)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -25.38 (2.66) | -33.47 (2.69) | -36.89 (2.71) | -49.38 (2.70) | -48.36 (2.64) | -8.35 (2.72)

14. Secondary Outcome: Change From Baseline in C- Reactive Protein (CRP) (mg/L)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Change = value at observation minus value at baseline.
Time Frame: Baseline, Week 2, 4, 8 and 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
mg/L
  Week 2 (n=53, 53, 51, 52, 54, 52) | -5.69 (2.24) | -16.61 (2.24) | -17.32 (2.29) | -22.50 (2.26) | -24.95 (2.22) | 1.02 (2.26)
  Week 4 (n=52, 51, 51, 52, 52, 52) | -5.56 (2.25) | -16.26 (2.27) | -22.20 (2.29) | -24.47 (2.26) | -24.59 (2.25) | 0.59 (2.26)
  Week 8 (n=51, 51, 51, 52, 52, 50) | -9.79 (2.27) | -16.71 (2.27) | -23.80 (2.29) | -23.56 (2.26) | -26.03 (2.25) | 5.27 (2.29)
  Week 12 (n=51, 49, 50, 49, 52, 48) | -8.88 (2.27) | -18.34 (2.30) | -23.97 (2.30) | -25.11 (2.30) | -26.14 (2.25) | 8.22 (2.32)

15. Secondary Outcome: Area Under Curve (AUC) for Change From Baseline in American College of Rheumatology-N (ACR-N)
Description: ACR-N = calculated for each participant by taking lowest percentage improvement in (1) swollen joint count or (2) tender joint count or (3) the median of remaining 5 components of ACR response (participant's assessment of disease activity; participant's global assessment of pain; physician's assessment of disease activity; participant's assessment of physical function; an acute phase reactant value - CRP). Negative numbers indicate worsening. The AUC for ACR-N is measure of the area under the curve of the mean change from baseline in ACR-N. The trapezoidal rule was used to compute AUC.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 54 | 52
units on a scale | 498.47 (341.96) | 1876.4 (341.96) | 2573.0 (345.23) | 3887.4 (341.96) | 3628.9 (338.78) | -2415 (345.23)

16. Secondary Outcome: Change From Baseline in Euro Quality of Life (EQ-5D)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state. Change = score at Week 12 minus score at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 0.10 (0.03) | 0.21 (0.03) | 0.28 (0.03) | 0.33 (0.03) | 0.33 (0.03) | -0.04 (0.03)

17. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Physical Functioning Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
  Change = score at Week 12 minus score at baseline.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 2.62 (1.09) | 6.23 (1.11) | 5.83 (1.13) | 9.59 (1.11) | 8.61 (1.08) | -2.53 (1.12)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Role-Physical Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.15 (1.18) | 4.42 (1.20) | 6.17 (1.21) | 8.91 (1.20) | 7.77 (1.17) | -0.72 (1.22)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Bodily Pain Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 5.94 (1.08) | 7.81 (1.10) | 9.74 (1.11) | 12.58 (1.10) | 13.90 (1.07) | 0.27 (1.12)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -General Health Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 2.12 (0.84) | 4.76 (0.86) | 5.37 (0.86) | 7.57 (0.86) | 7.61 (0.83) | 0.16 (0.87)

21. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Vitality Domain
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
  Change =score at Week 12 minus score at baseline
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- CP-690,550 5 mg BID: Participants were administered 5 mg of CP-690,550 orally twice daily for 12 weeks.
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg BID | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.67 (0.74) | 6.11 (0.76) | 6.58 (0.77) | 11.98 (0.77) | 9.49 (0.74) | 3.38 (0.79)

22. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Social Functioning Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 2.22 (1.21) | 4.88 (1.24) | 4.65 (1.24) | 4.56 (1.24) | 7.62 (1.20) | -0.67 (1.25)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Role-Emotional Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.83 (1.41) | 4.20 (1.44) | 5.64 (1.44) | 7.99 (1.44) | 6.42 (1.40) | -1.50 (1.47)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) -Mental Health Domain
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.29 (1.29) | 5.02 (1.32) | 8.62 (1.32) | 7.64 (1.32) | 6.27 (1.28) | 0.59 (1.34)

25. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) - Physical Component Summary (PCS)
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.27 (0.86) | 6.03 (0.88) | 6.22 (0.89) | 10.25 (0.88) | 10.27 (0.85) | -1.04 (0.89)

26. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) - Mental Component Summary (MCS)
Description: as for outcome 17
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Number analyzed (Participants) | 51 | 49 | 50 | 49 | 52 | 48
Units on a scale | 3.00 (1.27) | 3.99 (1.30) | 7.09 (1.30) | 6.15 (1.30) | 5.52 (1.26) | 0.15 (1.32)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 1 mg | CP-690,550 3 mg | CP-690,550 5 mg | CP-690,550 10 mg | CP-690,550 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 3/53 | 2/52 | 2/53 | 1/54 | 1/52
Other Adverse Events (participants affected / at risk) | 14/53 | 16/53 | 19/52 | 22/53 | 22/54 | 16/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=53) | CP-690,550 3 mg (N=53) | CP-690,550 5 mg (N=52) | CP-690,550 10 mg (N=53) | CP-690,550 15 mg (N=54) | Placebo (N=52)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid vasculitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 1 mg (N=53) | CP-690,550 3 mg (N=53) | CP-690,550 5 mg (N=52) | CP-690,550 10 mg (N=53) | CP-690,550 15 mg (N=54) | Placebo (N=52)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 4 | 6 | 3 | 8 | 6
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3
Blood cholesterol increased (Investigations) | 0 | 1 | 1 | 1 | 2 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 1 | 6 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 6 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 3 | 2 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.